CLINICAL TRIAL: NCT06112444
Title: Validity And Reliability Study Of The Turkish Version Of Short Western Ontario Rotator Cuff Index
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Selda Başar, Professor in University, Gazi University
Other Study IDs: 2023-1070
Record Dates: First submitted 2023-10-19; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Rotator Cuff Injuries
Keywords: validity of results; reliability of results
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: scale — The scale of Short Western Ontario Rotator Cuff İndex

SUMMARY:
The purpose of this study is to examine the psychometric properties of a Turkish shortened version of the Western Ontario Rotator Cuff Index (SHORTWORC).

DETAILED DESCRIPTION:
Many of the musculoskeletal diseases that doctors treat every day affect both quality of life and functionality. Rotator Cuff diseases are highly prevalent shoulder disorders associated with pain and functional limitations. Thus, surveys measuring treatment outcomes and activity limitations have become important in clinical research. Such scales can be time consuming or impractical for the patient, depending on the areas they evaluate. For this reason, the development of scales focusing on specific areas facilitates evaluations in the clinical environment. The purpose of this study is to examine the psychometric properties the Turkish SHORTWORC index, which is designed to focus on a single parameter.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-64
* the presence of rotator cuff pathology requiring surgical treatment

Exclusion Criteria:

* Chronic inflammatory diseases
* cervical spine radiculopathy
* different structural shoulder problems in the last three months
* previous surgery and associated additional pathologies requiring stabilization or other major *surgery such as superior labral repair
* any history of systemic disease
* being an athlete

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: İndividuals diagnosed with Rotator cuff disease by a specialist in Gazi University Faculty of Medicine Orthopedics and Traumatology Polyclinic constitute the sample of the study.
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Short Western Ontario Rotator Cuff Index | First Day
  The scale of Short Western Ontario Rotator Cuff Index is a disease-spesific index designed to evaluate activity limitations in patient with rotator cuff disorders. It is an abbreviated version of Western Ontario Rotator Cuff Index (WORC). İt has 7 items that access only 1 domain , the activity limitations. Patients rate their function on a scale from 0, meaning no difficulty, to 100, meaning extreme difficulty. The percentage scores for the Short-WORC are obtained by subtracting the total score from 700, dividing by 700, and multiplying by 100, resulting in a total percentage score varying from 0 to 100.,
Constant-Murley score (CMS) | First Day
  The Constant-Murley score (CMS) is a 100-points scale composed of a number of individual parameter. These parameters define the level of pain and the ability to carry out the normal daily activities of the patient. The Constant-Murley score was introduced to determine the functionality after the treatment of a shoulder injury.
American Shoulder and Elbow Surgeons Shoulder Score (ASES) | First Day
  The ASES is a 100-point scale that consists of two dimensions: pain and activities of daily living. There is one pain scale worth 50 points and ten activities of daily living worth 50 points. İt has been also reported to be reliable and valid in patients ,with upper extremity, shoulder or rotator cuff pathology.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No